CLINICAL TRIAL: NCT03311776
Title: BIOmarkers in Patients With PAncreatic Cancer (BIOPAC) - Can They Provide New Information of the Disease and Improve Diagnosis and Prognosis of the Patients?
Brief Title: BIOmarkers in Patients With Pancreatic Cancer ("BIOPAC")
Acronym: BIOPAC
Status: Recruiting | Type: Observational
Sponsor: Inna Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Inna Chen, MD, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: GI 0815
Record Dates: First submitted 2017-10-06; First posted 2017-10-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Biomarkers; Biobank; Diagnostic biomarkers; Predictive biomarkers; Prognostic biomarkers
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and tissue from primary tumor and/or metastasis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
No validated biomarkers to identify PC at an early stage and to predict treatment outcomes in the individual patient exist. The objective of the present study is to find diagnostic, prognostic and predictive biomarkers.

DETAILED DESCRIPTION:
The overall survival of patients with pancreatic cancer (PC) is dismal and has only improved slightly during the last decades primarily due to combination chemotherapy. Early detection of PC is difficult and less than 25% of all PC patients are operated. No validated biomarkers to identify PC at an early stage and to predict treatment outcomes in the individual patient exist. The objective of the present study is to find diagnostic, prognostic and predictive biomarkers, which can be used to 1) diagnose PC early in the disease course with high specificity and sensitivity, 2) improve prognostication, or 3) predict and monitor treatment effectiveness and tolerability for the individual patient.

BIOPAC is an observational and translational open cohort study with prospective collection of biological materials and clinical data in patients with PC treated in routine care and also patients who were suspicious for malignancy in the pancreas but then operated without evidence of malignancy. Patients contribute with blood samples (i.e. serum, EDTA plasma and buffy coat, and blood in PAXgeneRNA tubes) before operation or start of adjuvant or palliative chemotherapy and during treatment with blood sampling before 2. cycle of chemotherapy and longitudinally every time of CT scan until disease progression. This schedule is repeated if patients are treated with subsequent lines of chemotherapy. The patients are followed until death. Demographics, disease characteristics, comorbidities and lifestyle factors are registered at inclusion; weight and performance status at each treatment cycle; routine blood tests (i.e. haematology, creatinine, liver enzymes, bilirubin, carbohydrate antigen 19-9, C-reactive protein); type of operation; types of chemotherapy and number of cycles given; date of disease recurrence in operated patients; date of disease progression for each line of chemotherapy; and date of death. Biomarker analyses will include a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins and metabolites. Data will be analysed using appropriate methods and statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically verified PC (ductal adenocarcinoma) or ampullary adenocarcinoma in a resected specimen; or histopathological confirmation of carcinoma in patients not undergoing surgery in the setting of clinical and radiological characteristics which, together with the pathology, are consistent with a diagnosis of PC independently of stage

Exclusion Criteria:

• None

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with localized, locally advanced or metastatic PC treated in routine care in six hospitals in Denmark as well as operated patients who were suspicious for PC but without evidence of cancer in histology.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-07-03 (Actual); Primary Completion 2035-07-02 (Estimated); Study Completion 2035-07-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic biomarkers | baseline
  Biomarker analyses include, but are not limited to a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins and metabolites.
Prognostic biomarkers | baseline and through study completion, an average of 1 year
  Biomarker analyses include, but are not limited to a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins and metabolites.
Predictive biomarkers | baseline and through study completion, an average of 1 year
  Biomarker analyses include, but are not limited to a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins and metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev & Gentofte Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Pedersen RS, Nissen NI, Jensen C, Thorlacius-Ussing J, Manon-Jensen T, Olesen ML, Langholm LL, Diab HMH, Jorgensen LN, Hansen CP, Chen IM, Johansen JS, Karsdal MA, Willumsen N. Plasma Kallikrein-Activated TGF-beta Is Prognostic for Poor Overall Survival in Patients with Pancreatic Ductal Adenocarcinoma and Associates with Increased Fibrogenesis. Biomolecules. 2022 Sep 17;12(9):1315. doi: 10.3390/biom12091315. PMID 36139154
- [Derived] Nissen NI, Kehlet S, Johansen AZ, Chen IM, Karsdal M, Johansen JS, Diab HMH, Jorgensen LN, Sun S, Manon-Jensen T, He Y, Langholm L, Willumsen N. Noninvasive prognostic biomarker potential of quantifying the propeptides of Type XI collagen alpha-1 chain (PRO-C11) in patients with pancreatic ductal adenocarcinoma. Int J Cancer. 2021 Jul 1;149(1):228-238. doi: 10.1002/ijc.33551. Epub 2021 Mar 22. PMID 33687786
- [Derived] Rasmussen LS, Yilmaz MK, Falkmer UG, Poulsen LO, Bogsted M, Christensen HS, Bojesen SE, Jensen BV, Chen IM, Johansen AZ, Hansen CP, Hasselby JP, Hollander N, Nielsen SE, Andersen F, Bjerregaard JK, Pfeiffer P, Johansen JS. Pre-treatment serum vitamin D deficiency is associated with increased inflammatory biomarkers and short overall survival in patients with pancreatic cancer. Eur J Cancer. 2021 Feb;144:72-80. doi: 10.1016/j.ejca.2020.10.038. Epub 2020 Dec 17. PMID 33341448
- [Derived] Chen IM, Willumsen N, Dehlendorff C, Johansen AZ, Jensen BV, Hansen CP, Hasselby JP, Bojesen SE, Pfeiffer P, Nielsen SE, Hollander NH, Yilmaz MK, Karsdal M, Johansen JS. Clinical value of serum hyaluronan and propeptide of type III collagen in patients with pancreatic cancer. Int J Cancer. 2020 May 15;146(10):2913-2922. doi: 10.1002/ijc.32751. Epub 2019 Nov 11. PMID 31642523
- [Derived] Mellby LD, Nyberg AP, Johansen JS, Wingren C, Nordestgaard BG, Bojesen SE, Mitchell BL, Sheppard BC, Sears RC, Borrebaeck CAK. Serum Biomarker Signature-Based Liquid Biopsy for Diagnosis of Early-Stage Pancreatic Cancer. J Clin Oncol. 2018 Oct 1;36(28):2887-2894. doi: 10.1200/JCO.2017.77.6658. Epub 2018 Aug 14. PMID 30106639